CLINICAL TRIAL: NCT06510751
Title: Evaluation of the Levels of Calcitonin Gene-related Peptide and Substance P in Patients With Post-operative Meningitis
Brief Title: Evaluation of the Levels of Calcitonin Gene-related Peptide and Substance P
Status: Recruiting | Type: Observational
Sponsor: Melike Cengiz (Other)
Responsible Party: Sponsor-Investigator, Melike Cengiz, MD,Professor Doctor, Akdeniz University
Organization: Akdeniz University (Other)
Other Study IDs: Akdeniz U. Faculty Medicine
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Meningitis; Diagnosis; Prognosis
Keywords: Postoperative meningitis; Calcitonin gene-related peptide; Substance P
MeSH Terms: conditions — Meningitis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 16 Months
Biospecimen Retention: Samples Without DNA — Cerebrospinal fluid Serum plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Postoperative meningitis mortality: Patients with postoperative meningitis and mortality in the intensive care unit.
  Interventions: Other: CGRP level
- Postoperative meningitis survival: Patients who developed postoperative meningitis and were discharged from the intensive care unit.
  Interventions: Other: CGRP level

INTERVENTIONS:
Other: CGRP level — CGRP and substance P levels will be analysed by ELISA method in CSF and blood materials.
  Other Names: Substans P level

SUMMARY:
In cases of meningitis caused by external ventricular catheters (EVDs), which are the most commonly placed intracranial catheters that can lead to central nervous system infection through contamination/colonisation, the diagnosis may not be differentiated by either clinical signs and symptoms or conventional cerebrospinal fluid (CSF) tests. Therefore, due to the limitations in diagnosis and prognostic prediction of EVD-induced meningitis and the high mortality/morbidity rates of the disease, markers with high sensitivity and specificity in post-operative meningitis are needed. Calcitonin gene-related peptide (CGRP), a neuropeptide, has been shown to increase when C or Aδ sensory fibres are damaged or in the presence of inflammation in tissues adjacent to the fibres. CGRP is localised in nociceptive nerve terminals together with another neuropeptide, substance P, which has similar biological effects. There are very few studies investigating how CGRP levels in CSF and serum change in bacterial meningitis. Although it is thought that nociception and neuroimmune interactions affect meningeal antibacterial host defence, that nociceptors signal via CGRP to meningeal immune cells during infection, and that this neuroimmune axis exacerbates bacterial meningitis by weakening host defence, it is not yet clear how CGRP and substance P levels affect disease prognosis. This study will evaluate the utility of CGRP and substance P levels as biomarkers to assess diagnosis and treatment response in patients with post-operative meningitis followed in the intensive care unit.

DETAILED DESCRIPTION:
Adult patients (18 years of age and older) with suspected CSF drainage system-related meningitis who are followed up in the Intensive Care Unit will be included in the study. Blood and CSF samples taken during routine clinical practice (before the development of meningitis symptoms, just before the first dose of antibiotherapy on the first day of meningitis symptoms, after the last dose of antibiotherapy on the 3rd day of antibiotherapy), CSF smear, CSF culture and CSF direct examination, CSF biochemistry parameters will be studied, and the materials will be taken into tubes containing aprotinin (proteinase inhibitor) to study CGRP and substance P levels in blood and CSF materials to be destroyed. CGRP and substance P levels will be analysed by ELISA method. Among the clinical parameters, the patient's state of consciousness (Glasgow coma scale), fever response, vasoactive drug requirement, organ failure, sepsis and septic shock status, SOFA and APACHE II scores will be recorded. Laboratory parameters available in routine clinical practice (haemogram, biochemical tests, microbiological growths, infection parameters), radiographic examination findings (computed brain tomography, brain magnetic resonance imaging), intensive care unit length of stay and intensive care unit outcomes (survival/mortality) will also be recorded for use in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over
* Patients followed up in the intensive care unit with suspected meningitis

Exclusion Criteria:

* Patients under 18 years of age
* Patients with suspected meningitis in the intensive care unit who have not undergone neurosurgical operation and do not have CSF drainage catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postoperative meningitis patients
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Diagnosis | 16 months
  The role of CGRP and substance P levels in blood and CSF samples in the diagnosis of postoperative meningitis

SECONDARY OUTCOMES:
Prognosis | 16 months
  The role of CGRP and substance P levels in blood and CSF samples in the evaluation of postoperative meningitis treatment response and prediction of patient prognosis

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University School of Medicine, Department of Anesthesiology and Intensive Care, Turkey, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No